CLINICAL TRIAL: NCT02401282
Title: Attention and Social Behavior in Children
Acronym: BRAINS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Penn State University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Koraly E. Perez-Edgar, Associate Professor of Psychology, Penn State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 5R01MH094633-04 (NIH); 5R01MH094633-04 (NIH)
Record Dates: First submitted 2015-03-24; First posted 2015-03-27 (Estimated); Last update posted 2018-01-16 (Actual); Status verified 2018-01

CONDITIONS: Anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- ABM (Experimental): Attention bias modification
  Interventions: Behavioral: Attention Bias Modification
- Placebo (Placebo Comparator): Dot-probe task
  Interventions: Behavioral: Dot-probe task

INTERVENTIONS:
Behavioral: Attention Bias Modification — This is a modification of the dot-probe task (placebo task) designed to train attention away from threat
  Arms: ABM
Behavioral: Dot-probe task — This is the active control placebo condition that simply measures levels of attention to threat
  Arms: Placebo

SUMMARY:
This study examines the way attention may be linked to temperamental risk for anxiety, social behavior and brain processes. The study aims to see if temperamentally at risk youth display an attention bias towards threat, and if anxiety symptoms can be reduced through attentional bias modification training.

ELIGIBILITY:
Inclusion Criteria:

* 9-12 year olds who do not meet exclusionary criteria (split into groups based on high and low temperamental shyness)

Exclusion Criteria:

* presence or permanent metal orthodontics or implanted metal devices
* severe psychiatric diagnosis
* IQ under 70 as assessed by the WISC

Ages: 9 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 251 (Actual)
Dates: Start 2011-12; Primary Completion 2016-12-17 (Actual); Study Completion 2016-12-17 (Actual)

PRIMARY OUTCOMES:
Anxiety Symptoms | 8 weeks
  parent and child report of child's anxiety symptoms
Attention bias levels | 8 weeks
  performance on computerized attention task
Electrophysiological and neural correlates of attention bias | 8 weeks
  EEG and fMRI measures

CONTACTS AND LOCATIONS:
Locations (1):
- Penn State University Child Study Center, University Park, Pennsylvania, United States

REFERENCES:
- [Background] LoBue V, Perez-Edgar K. Sensitivity to social and non-social threats in temperamentally shy children at-risk for anxiety. Dev Sci. 2014 Mar;17(2):239-47. doi: 10.1111/desc.12110. Epub 2013 Nov 28. PMID 24283271
- [Background] McDermott JM, Perez-Edgar K, Henderson HA, Chronis-Tuscano A, Pine DS, Fox NA. A history of childhood behavioral inhibition and enhanced response monitoring in adolescence are linked to clinical anxiety. Biol Psychiatry. 2009 Mar 1;65(5):445-8. doi: 10.1016/j.biopsych.2008.10.043. Epub 2008 Dec 24. PMID 19108817
- [Background] Perez-Edgar K, McDermott JN, Korelitz K, Degnan KA, Curby TW, Pine DS, Fox NA. Patterns of sustained attention in infancy shape the developmental trajectory of social behavior from toddlerhood through adolescence. Dev Psychol. 2010 Nov;46(6):1723-30. doi: 10.1037/a0021064. PMID 20873921
- [Background] Perez-Edgar K, Reeb-Sutherland BC, McDermott JM, White LK, Henderson HA, Degnan KA, Hane AA, Pine DS, Fox NA. Attention biases to threat link behavioral inhibition to social withdrawal over time in very young children. J Abnorm Child Psychol. 2011 Aug;39(6):885-95. doi: 10.1007/s10802-011-9495-5. PMID 21318555
- [Background] Perez-Edgar K, Roberson-Nay R, Hardin MG, Poeth K, Guyer AE, Nelson EE, McClure EB, Henderson HA, Fox NA, Pine DS, Ernst M. Attention alters neural responses to evocative faces in behaviorally inhibited adolescents. Neuroimage. 2007 May 1;35(4):1538-46. doi: 10.1016/j.neuroimage.2007.02.006. Epub 2007 Feb 15. PMID 17376704
- [Background] Williams LR, Degnan KA, Perez-Edgar KE, Henderson HA, Rubin KH, Pine DS, Steinberg L, Fox NA. Impact of behavioral inhibition and parenting style on internalizing and externalizing problems from early childhood through adolescence. J Abnorm Child Psychol. 2009 Nov;37(8):1063-75. doi: 10.1007/s10802-009-9331-3. PMID 19521761
- [Derived] Liu P, Taber-Thomas BC, Fu X, Perez-Edgar KE. Biobehavioral Markers of Attention Bias Modification in Temperamental Risk for Anxiety: A Randomized Control Trial. J Am Acad Child Adolesc Psychiatry. 2018 Feb;57(2):103-110. doi: 10.1016/j.jaac.2017.11.016. Epub 2017 Nov 28. PMID 29413142